CLINICAL TRIAL: NCT02397148
Title: Assessment of the Morphological Concordance Between CT and Cone Beam in Sinus Imagery
Acronym: COSINUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13 147 03; 2013-A00736-39 (Registry Identifier: ANSM)
Record Dates: First submitted 2015-03-04; First posted 2015-03-24 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2016-10

CONDITIONS: Sinonasal Pathologies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients with sinonasal pathology (Experimental): Computed Tomography Cone Beam Computed Tomography
  Interventions: Radiation: Computed Tomography; Radiation: Cone Beam Computed Tomography

INTERVENTIONS:
Radiation: Computed Tomography — imagery with ionizing radiation
Radiation: Cone Beam Computed Tomography — imagery with ionizing radiation

SUMMARY:
This study compares the morphological concordance between CT (computed tomography) and cone beam in sinus on 26 validated items. CT and cone beam is performed on each patient. Performances of these two imagery technics seem to be closed. Nevertheless, the exposure of the ionizing radiations is lower with the cone beam.

ELIGIBILITY:
Inclusion Criteria:

* man or woman older than 18 years old
* patient affected by sinonasal pathology : who show one or more of the following functional sign : anosmia, pain with sinusal origin (frontal headache, lower-orbital throbbing pain increased in anteflexion, chronic unexplained headache), nasal blockage, runny nose, epistaxis requiring the realisation of a sinus imagery overview.

Exclusion Criteria:

* Deprivation of liberty by administrative or legal decision
* patients under 18 years old
* Patients in emergency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
intraclass correlation coefficient | 1 day
  Assessment of the morphological concordance between the CT and the Cone Beam in the sinus imagery with 26 validated items.

SECONDARY OUTCOMES:
morphological concordance between cone beam and CT | 1 day
  Assessment of the morphological concordance between the CT and the Cone Beam in the sinus imagery with these 26 items assessed separately
reproductibility INTER-OBSERVER | 1 day
  The reproducibility of the measurement between the two neuroradiologists will be assessed by intraclass correlation coefficient, based on 26 benchmarks of primary endpoint. Similarly inter-observer reproducibility will be assessed for the 36 specific criteria
dosimetry | 1 day
  Assessment of the dosimetry CT/ Cone Beam
Diagnosis concordance radio-endoscopic and radio-surgical | 1 day
  Radio-endoscopic surgical concordance and radio will be estimated by calculating the proportion of concordant diagnoses between the radiological evaluation and cone beam scanner and endoscopic evaluation obtained at the first nasal endoscopy and radiological evaluation between the scanner and cone beam and intraoperative assessment in case of surgery. The investigators then compare the radio-endoscopic surgical concordance and radio and the cone beam scanner.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien VERGEZ, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- VERGEZ, Toulouse, France

REFERENCES:
- [Result] Demeslay J, Vergez S, Serrano E, Chaynes P, Cantet P, Chaput B, de Bonnecaze G. Morphological concordance between CBCT and MDCT: a paranasal sinus-imaging anatomical study. Surg Radiol Anat. 2016 Jan;38(1):71-8. doi: 10.1007/s00276-015-1509-5. Epub 2015 Aug 4. PMID 26239897